CLINICAL TRIAL: NCT06865352
Title: Phase I/IIa Clinical Trial on the Safety and Preliminary Efficacy of Donor-derived Anti-leukemia Cytotoxic T Lymphocytes for the Prevention of Leukemia Relapse in Children Given Haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: Safety and Preliminary Efficacy of Donor-derived Anti-leukemia Cytotoxic T Lymphocytes for the Prevention of Leukemia Relapse in Children Given Haploidentical Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Marco Zecca, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Leuk-CTL-001
Record Dates: First submitted 2025-02-28; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Acute Lymphoblastic Leukemia ALL; Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients cohort (Experimental): single-arm study: patients receive leukemia-specific CTLs
  Interventions: Biological: HSCT donor leukemia-specific cytotoxic T-cells

INTERVENTIONS:
Biological: HSCT donor leukemia-specific cytotoxic T-cells — donor T-cells stimulated with patient leukemia blasts

SUMMARY:
The prognosis for children affected by acute leukemia and transplanted in an advanced disease stage, in the presence of MRD or with unfavorable cytogenetic abnormalities, is still poor. Optimizing post-transplant management to maintain durable remission represents the greatest challenge to improve the outcome of pediatric patients with acute leukemia given an allogeneic HSCT.

The pivotal therapeutic role of immunity against acute leukemia has been highlighted by the immunological effect of donor T cells (GVL) observed following allogeneic HSCT, which is considered the only curative strategy for this type of cancer. Moreover, circulating leukemia-specific CTLs have been detected in patients with different forms of acute leukemia, and the presence of these specific T-cell responses in peripheral blood and bone marrow samples of leukemic patients has been associated with improved disease control and longer survival. This body of data suggests that immunological interventions could have an effect in preventing relapse and improving transplant outcome.

Unmanipulated donor lymphocyte infusion (DLI) is used after stem cell transplantation to treat and prevent relapse, to prevent infections and to establish full donor chimerism. However, an expected side effect of the presence of mature T cells is the potential occurrence of acute GvHD. Evidence has emerged that escalating DLI has achieved higher clinical response rates with lower GvHD occurrence. Optimization of DLI dose and schedule as well as strategies of donor T-cell manipulation may lead to the consistent ability to separate GvHD from GvL activity and improve the safety of DLI treatment. One way to manipulate donor lymphocytes to reduce GVHD is leukemia antigen stimulation, in order to increase antileukemia activity while reducing the number of alloreactive T cells by specific culture.

The aim of this study is to enhance the GVL effect, and reduce the rate of post-transplant relapse, with preventive post-HSCT infusions of donor anti-leukemia CTLs specifically directed to patient's leukemic blasts. The leukemia-reactive CTLs obtained by stimulation with patients' leukemia blasts are specific for each individual blast signature, and, due to their physiological recognition and effector mechanism through their natural T cell receptor, exert leukemia-specific killing with less severe adverse reactions than CAR-T cells. Moreover, due to their potential to recognize multiple leukemia-associated antigens present on the blast surface, they should be less prone to immune evasion strategies exerted by leukemic stem cells. Additionally, the risk of GVHD should be reduced by the culture procedure, which decreases the number of alloreactive T cells. For the reasons stated, the use of these T cells after HSCT in a highly personalized approach may be a safer and more efficient option than unmanipulated donor lymphocyte infusions (DLIs) to prevent leukemia relapse after HSCT.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Age ≤ 18 years and ≥ 1 months
2. Life expectancy > 12 weeks
3. Patients affected by life-threatening acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML) with high risk of relapse after HSCT, namely:

   Patients affected by ALL:
   * in first morphological remission but with a positive minimal residual disease ≥ 1 x 10-3 before HSCT;
   * in second morphological remission after a high-risk relapse (patients belonging to the S3-S4 BFM risk group), independently of the level of minimal residual disease;
   * in second morphological remission with any positivity of minimal residual disease before HSCT;
   * in third or subsequent morphological remission, independently of the level of minimal residual disease;
   * patients not in morphological remission at time of HSCT.

   Patients affected by AML:
   * in first morphological remission and with a flow cytometry MRD at the end of induction therapy ≥ 0.1%;
   * in first morphological remission and with high-risk disease according to cytogenetics aberrations;
   * in first morphological remission after a primary induction failure;
   * in second morphological remission;
   * in third or subsequent morphological remission;
   * patients not in morphological remission at time of HSCT.
4. Pre-HSCT Lansky / Karnofsky score ≥ 40%.
5. HIV negativity.
6. Written informed consent signed by the parents or legal guardians (in case of patients < 18 years) or by the patients (in the case of patients = 18 years).

Patient Exclusion Criteria:

1. Ongoing active ≥ grade II acute GvHD or chronic extensive GvHD due to a previous allograft
2. Current clinically active infectious disease (including positive HIV serology or viral RNA)
3. Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or left ventricular ejection fraction <40%)
4. Liver dysfunction (AST/ALT ≥ 3 times institutional upper limit normal value -ULN- or bilirubine > 3 times ULN)
5. Renal dysfunction: serum creatinine > 1.5 times ULN or calculated creatinine clearance < 60 ml/min/1.73 m2
6. End stage irreversible multi-system organ failure.
7. Other active malignancy.
8. Pregnant or breast feeding female patient
9. Lack of parents'/guardian's written informed consent for minors or lack of written informed consent for patients aged 18 y.

Donor inclusion criteria:

Eligible donors are the HSCT donors, i.e. HLA-haploidentical relative, including but not limited to biological parents, siblings, or half-siblings. Matching will be determined by class I and class II DNA typing.

1. Age between 18 and 65 years.
2. The donor should be sufficiently healthy not to be at increased risk from the leukapheresis procedure.
3. Donors must meet the selection criteria as defined by the European Directive 2006/17/CE) and according to the FACT-JACIE International Standards and local regulations for donor selection.
4. Donor must have adequate peripheral venous access for leukapheresis or must agree to placement of a central venous catheter.
5. Signed informed consent.

Donor exclusion criteria:

1. Evidence of active infection (including urinary tract infection, or upper respiratory tract infection) or viral hepatitis exposure (on screening), unless HBs Ab+ and HBV DNA negative.
2. Factors which place the donor at increased risk for complications from leukapheresis (e.g. autoimmune disease, symptomatic sickle cell trait, symptomatic coronary artery disease requiring therapy, previous thrombotic events).
3. Pregnancy or breastfeeding female donor.
4. Lack of written informed consent.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-13 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Safety evaluated as the incidence of acute GVHD | during the study and end of study
  Acute GVHD will be diagnosed and graded according to the NIH criteria. Grade II-IV acute GVHD will be expressedas cumulative incidence (CI) considering disease relapse and death in remission without GVHD as competing events. A CI of acute GVHD ≤ 25% will be considered as acceptable treatment toxicity.

SECONDARY OUTCOMES:
Relapse (REL) | Relapse will be calculated at 3, 6, 9, 12 18 and 24 months after HSCT
  REL, defined as the time from HSCT to the date of disease relapse will be expressed as cumulative incidence (CI) considering death in remission as a competing event. The CI of REL in treated patients will be compared with that of recipients of haplo-HSCT with the same disease characteristics and prognosis, give conventional infusions of unmanipulated, donor-derived T lymphocytes (DLI). Preliminary efficacy of the treatment will be a CI of REL ≤ of the CI of REL observed in the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Ematologia 2 - Oncoematologia Pediatrica, Pavia, Pavia, Italy

REFERENCES:
- [Derived] Montagna D, Comoli P, Tanzi M, Montini E, Moretta A, Taurino G, Boghen S, Panigari A, Mina T, Giorgiani G, Del Fante C, Perotti C, Zecca M. Phase I/II clinical trial on the safety and preliminary efficacy of donor-derived anti-leukemia cytotoxic T lymphocytes for the prevention of leukemia relapse in children given haploidentical hematopoietic stem cell transplantation: study rational and design. Front Immunol. 2025 Jun 6;16:1601961. doi: 10.3389/fimmu.2025.1601961. eCollection 2025. PMID 40547030